CLINICAL TRIAL: NCT06833307
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating Efficacy and Safety of SHR-1314 in the Treatment of Pediatric Patients of Age 6 to <18 Years With Moderate to Severe Plaque Psoriasis
Brief Title: The Efficacy and Safety of SHR-1314 in the Treatment of Pediatric Patients of Age 6 to <18 Years With Moderate to Severe Plaque Psoriasis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1314-307
Record Dates: First submitted 2025-02-11; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Children and Adolescents Aged 6 to 18 With Moderate-to-Severe Plaque Psoriasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1314 (Experimental)
  Interventions: Drug: SHR-1314

INTERVENTIONS:
Drug: SHR-1314 — SHR-1314: dose 1 SHR-1314:dose 2 SHR-1314:dose 3

SUMMARY:
The purpose of this study is to assess efficacy, safety of subcutaneous SHR-1314 in pediatric patients of age 6 to <18 years with moderate-to-Severe plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. between 6 and 18years of age at time of screening.
2. Chronic plaque-type psoriasis present for at least 6 months and diagnosed before randomization.
3. Moderate to severe psoriasis as defined at Baseline/ randomization by:

PASI score of 12 or greater, and sPGA score of 3 or greater (based on a static scale of 0 - 5), and Body Surface Area (BSA) affected by plaque psoriasis of 10% or greater.

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and guttate psoriasis) at Screening or Baseline/randomization.
2. Drug-induced psoriasis.
3. Had a clinically significant flare of psoriasis during the 12 weeks prior to baseline (Week 0).
4. Presence of other skin conditions (e.g. skin infections, seborrheic dermatitis) that in the judgement of the Investigator could interfere with assessment of psoriasis.
5. History of inflammatory bowel disease or have other ongoing active autoimmune diseases.
6. At screening, history or symptoms of malignancy of any organ system, treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
7. History of congestive heart failure (New York Heart Association [NYHA] functional classification ≥III), cerebro-cardiovascular events, or serious bleeding events at screening and / or randomization that in the judgement of the Investigator prevents the subject from participating in the study.
8. Active systemic infections (other than common cold) during the 4 weeks before randomization (e.g., hepatitis), or serious infections requiring hospitalization and/or intravenous injection of antibiotic treatment within eight weeks prior torandomization.
9. History of depression and/or suicidal ideation or any suicidal behavior based on an assessment with the Columbina Suicide Severity Rating Scale (C-SSRS) at screening and baseline (Posner K et al, 2011), The subjects will be exluded if any answer to question is "yes" in the questionnaire orare clinically judged by the investigator to be at risk for suicide.
10. All subjects will be tested for tuberculosis status using IGRA and X-ray test.
11. Have evidence of positive test for hepatitis B, hepatitis C antibody, or human immunodeficiency virus (HIV) antibodies.
12. Have a known allergy or hypersensitivity to any biologic therapy at screening that would pose an unacceptable risk to the subject if participating in this study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Safety assessment including adverse events at Week 16 | Week 16
PK parameters: Cmax at Week 12 | Week 12

SECONDARY OUTCOMES:
Percentage of subjects who achieve at least 75% improvement in PASI score (PASI 75) at Week 12 | Week 12
sPGA of 0 or 1 response at Week 12 | Week 12
Percentage of subjects who achieve at least 90% improvement in PASI score (PASI 90)at Week 12 | Week 12

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Capital Medical University Affiliated Children's Hospital, Beijing, Beijing Municipality
  - Shanghai Huashan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided